CLINICAL TRIAL: NCT06798311
Title: Reducing Disparities in Urinary Control Symptoms for Minority Women
Acronym: SUPPORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB24-1131; 5R01DK129849-04 (NIH)
Record Dates: First submitted 2025-01-22; First posted 2025-01-29 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Urinary Incontinence (UI); Lower Urinary Tract Symptoms (LUTS); Pelvic Floor Disorder
Keywords: cognitive behavioral therapy; self-directed; physical therapy; behavioral modifications; pelvic floor; home-based; health disparities
MeSH Terms: conditions — Urinary Incontinence; Lower Urinary Tract Symptoms; Pelvic Floor Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SUPPORT workbook (Experimental): All enrolled patients will be given access to the SUPPORT workbook (hard copy and PDF). The SUPPORT workbook contains a template for how pelvic floor physical therapy is delivered in the typical in-person setting with a combination of education, bladder re-training exercises, pelvic floor stretching and core strengthening. Patients also will be given access to a custom programmed GPT trained on the SUPPORT workbook and given instructions on empathetic communication techniques and assisting patients in performing the SUPPORT exercises as outlined in the program.
  Interventions: Behavioral: SUPPORT workbook

INTERVENTIONS:
Behavioral: SUPPORT workbook — The SUPPORT workbook contains a template for how pelvic floor physical therapy is delivered in the typical in-person setting with a combination of education, bladder re-training exercises, pelvic floor stretching and core strengthening. To aid in the demonstration of physical therapy exercises, the workbook includes QR-coded links to videos of a physical therapist performing the exercises in an ideal form. The videos include audio instruction to ensure that patients can learn the concepts in either visual, auditory or written form. The cognitive behavioral therapy (CBT) portion of the workbook is adapted from the standardized CBT protocol and includes short introductions and exercises pertaining to cognitive flexibility, behavioral activation and social support. The total time commitment for the program is 2-hours per week.
  Patients also will be given access to a custom programmed GPT trained on the SUPPORT workbook and given instructions on empathetic communication techniques.
  Other Names: cognitive behavior therapy

SUMMARY:
The study is designed to address the disparity in available conservative/behavioral treatments for UI/LUTS. The program was developed by experts from urogynecology, psychology, and physical therapy then modified based on focus group feedback from racially minoritized women. The study team created a patient-centered, culturally adapted, self-directed, 8-week, home-based module for women with LUTS/UI. The SUPPORT program combines multiple evidence-based conservative treatments for LUTS/UI including cognitive behavioral therapy, behavioral modifications, and home physical therapy exercise. Progression through the home-based program is supported by research staff. This prospective interventional study aims to evaluate the feasibility and acceptability of the SUPPORT program and its impact on patient-centered treatment outcomes, while enabling comparisons across race and ethnicity. This approach will provide a comprehensive understanding of how to effectively deliver self-management strategies for pelvic floor disorders.

At the start of the 8 week SUPPORT course participants will also be given access to a custom programmed GPT trained on the SUPPORT workbook and given instructions on empathetic communication techniques and assisting patients in performing the SUPPORT exercises as outlined in the program. At the end of 8 weeks patients will fill out a survey assessing the frequency of use and interactions with the LLM.

DETAILED DESCRIPTION:
Several recent large, population-based studies report that the prevalence of bothersome urinary incontinence (UI) and lower urinary tract symptoms (LUTS) ranges from 55-73%, and a woman's lifetime risk of surgery for pelvic floor disorders is 20%. In other words, one in every five women can expect to undergo surgery for UI or prolapse by age 80, underscoring the public health impact of these conditions. For perspective, a woman's lifetime risk of breast and lung cancer are 15% and 6%, respectively. Although the lifetime risk of UI/LUTS is significantly higher than that of breast cancer or lung cancer, UI/LUTS have not received the same level of attention by the public or the healthcare community, despite the severe consequences on quality of life. Women are often embarrassed to seek treatment and lack knowledge about how to manage these bothersome conditions. These barriers lead to reduced healthcare-seeking for these disorders, which further exacerbates the detrimental consequences for quality of life. Similarly, the study team recently found in a geographically diverse, population-based study that housing insecurity, unreliable transportation, housing insecurity, not having enough money to make ends meet, and percent federal poverty levels of 300% or less were associated with more LUTS and lower perceived bladder health.

Additionally, there are disparities in access to treatment for PFDs and inclusion in PFD research for racially minoritized women. One important disparity is the lack of access to evidence-based non-surgical options (e.g., diet and weight loss counseling, behavioral modification, physical therapy (PT), and cognitive behavioral therapy (CBT)) that should be recommended to most women because these treatments can treat multiple PFDs and restore quality of life without the need for more invasive approaches. These conservative interventions are often not offered to racially minoritized women due to poor access and coverage. Improving non-surgical treatment of bladder symptoms is crucial because treatments are complex and multidimensional; treating one symptom surgically can sometimes exacerbate other symptoms. Up to 6% of women who have surgery for stress urinary incontinence (SUI) will undergo a second surgery within 9 years. Women are also at increased risk for de novo urinary symptoms (urinary incontinence and urinary tract infection) after surgical interventions. Likewise, bladder symptoms lead to emotional distress (i.e., anxiety and depression), and in turn, emotional distress can exacerbate UI/LUTS. In order to prevent this cycle of cumulative symptoms and distress, environmental barriers to LUTS must be reduced, and publicly-insured women of low socio-economic status should be able to have the same access to non-surgical interventions as privately insured women.

Pelvic floor physical therapy (PFPT) is a well-established first-line treatment for UI/LUTS. A 2014 Cochrane Review, which included 21 trials with 1281 incontinent women, compared pelvic floor muscle exercises to sham or control treatments. Patients who performed pelvic floor muscle exercises were 17 times more likely to be cured or improved. Standard pelvic floor physical therapy, which combines behavioral retraining and manual muscle therapy, takes 8-12 sessions and requires insurance coverage, copays, travel, a significant time commitment, and effective communication with the therapist. Although some hospitals employ pelvic floor physical therapists, most operate within private practices and do not work with Medicaid or Medicare payers. Likely as a result of these disparities, prior studies have found that racially minoritized women are more likely to assume that surgery is the only treatment option for PFDs.

This study is designed to address the disparity in available conservative/behavioral treatments for UI/LUTS. The investigators created a patient-centered, culturally adapted, self-directed, 8-week, home-based module for women with LUTS/UI. The SUPPORT program combines multiple evidence-based conservative treatments for LUTS/UI, including cognitive behavioral therapy, behavioral modifications, and home physical therapy exercises. The program was developed by experts from urogynecology, psychology, and physical therapy, and then modified based on focus group feedback from racially minoritized women. The inclusion of women from all races and ethnicities in the study will allow for comparisons across groups, providing the fullest understanding of how to deliver effective self-management for pelvic floor disorders. Progression through the home-based program is supported by research staff. The aim of this prospective interventional study is to assess the feasibility and acceptability of the SUPPORT program and its impact on patient-centered treatment outcomes.

The SUPPORT workbook follows a template for how pelvic floor physical therapy is delivered in the typical in-person setting with a combination of education, bladder re-training exercises, pelvic floor stretching, and core strengthening. The educational topics were chosen by consensus among the clinical experts as the most common and important clinical contributors to UI/LUTS symptoms and common areas of patient misinformation.

To aid in the demonstration of physical therapy exercises, the workbook includes QR-coded links to videos of a physical therapist performing the exercises in an ideal form. The videos include audio instruction to ensure that patients can learn the concepts in either visual, auditory, or written form.

Recognizing the limited time that patients have to engage with this intervention and mimicking the time commitment of standard pelvic floor PT, the investigators aimed to have the program take no more than 2 hours per week. This time commitment is split between time dedicated to reading the chapter, time spent completing the physical therapy or cognitive behavioral therapy exercises on a daily basis, and the time spent engaging in physical activity of the patient's choosing. Patients are counseled that exercise is important to the program as it improves core strength, pelvic floor mobility, bowel motility, and behavioral activation while reducing anxiety.

The cognitive behavioral therapy (CBT) portion of the workbook is adapted from the standardized CBT protocol and includes short introductions and exercises pertaining to cognitive flexibility, behavioral activation, and social support.

Recent advances in artificial intelligence, particularly in the development of large language models (LLMs), have opened new possibilities in healthcare. The investigators also aim to explore the use of a customized LLM-based health coach to assist women participating in the SUPPORT program. By providing real-time support and guidance, the AI health coach could help overcome barriers to care and keep patients engaged in the treatment. This approach has the potential to enhance the effectiveness of self-management programs for pelvic floor disorders, making care more accessible and helping more women achieve better health outcomes.

Major goals of the study include:

Aim 1. To use a human-centered, iterative approach with qualitative interviews to create and adapt a self-managed CBT (SM-CBT) intervention along with a self-directed behavioral modification/PT (Home PT) program for women with UI/LUTS from all races and ethnicities, including those who are minority, low-income, and publicly insured.

Aim 2. To determine the efficacy of the SUPPORT intervention on UI/LUTS outcomes as well as patient acceptability and adherence.

Aim 3. To evaluate a large language model-based digital coach's ability to be integrated into a self-managed pelvic floor program.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to converse in English
* A response of at least "somewhat bothered" by urinary incontinence, urinary frequency or urgency on the UDI
* Willing to engage in conservative treatment of their UI/LUTS for 16 weeks

Exclusion Criteria:

* Anterior or posterior pelvic organ prolapse beyond the hymen or apical prolapse to the hymen
* Currently taking medications for their UI/LUTS or history of surgical intervention for UI
* Patients with abnormal PVR and positive urine culture at time of study entry
* History of recurrent UTIs
* History of mobility or neurologic disorders that would prevent ability to complete at home physical therapy
* Planning to start PT within the next 16 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Urinary Symptom Changes (UDI Subscale) | From enrollment to the end of treatment at 8 weeks
  To compare changes in urinary symptoms using the validated Urinary Distress Inventory (UDI) subscale of the Pelvic Floor Distress Inventory (PFDI) between baseline and 8-weeks (program completion) in patients undergoing the SUPPORT program. The Urinary Distress Inventory (UDI-6) is a validated 6-item questionnaire that assesses lower urinary tract symptoms, including incontinence, in women. The UDI-6 score is calculated by averaging the responses to each question (possible value 0 to 4), then multiplying that average by 25 to scale the score from 0 to 100. A higher score indicates greater distress.

SECONDARY OUTCOMES:
Urinary symptoms - UDI-6 (16 Weeks) | From enrollment to 16 weeks after SUPPORT program initiation
  To compare changes in urinary symptoms using the UDI between baseline and 16 weeks (2 months after program completion) after SUPPORT program initiation.
  The Urinary Distress Inventory (UDI-6) is a validated 6-item questionnaire that assesses lower urinary tract symptoms, including incontinence, in women. The UDI-6 score is calculated by averaging the responses to each question (possible value 0 to 4), then multiplying that average by 25 to scale the score from 0 to 100. A higher score indicates greater distress.
Urinary symptoms - LURN SI-10 (16 Weeks) | From enrollment to 16 weeks after SUPPORT program initiation
  To compare changes in urinary symptoms using the LURN SI-10 between baseline and 16 weeks (2 months after program completion) after SUPPORT program initiation.
  LURN Symptom Index-10 (LURN SI-10) were developed as patient-reported outcome measures to assess urinary symptoms in adult men and women. Higher scores indicate greater severity of LUTS. Scores on the LURN SI-10 range from 0 (least severe) to 38 (most severe).
Patient Global Impression of Improvement (PGI-I) | From enrollment to 16 weeks after SUPPORT program initiation
  To describe self-reported Patient Global Impression of Improvement (PGI-I) scores at 8 and 16 weeks after SUPPORT program initiation. The Patient global impression of improvement scale (PGI-I) is a single-item global rating of change scale that ask an individual patient to rate the severity of a specific condition. There are seven possible responses (scored 1-7): very much better, much better, a little better, no change, a little worse, much worse, and very much worse.
Pelvic Organ prolapse Distress Inventory and Colorectal-Anal distress Inventory subscales | From enrollment to 16 weeks after SUPPORT program initiation
  To compare changes in prolapse and bowel symptoms using the Pelvic Organ prolapse Distress Inventory 6 (POPDI-6) and Colorectal-Anal distress Inventory 8 (CRAD-8) at 8 and 16 weeks after SUPPORT program initiation. Both are subscales within the validated PFDI-20 questionnaire, used to assess the severity of symptoms related to pelvic organ prolapse and bowel dysfunction, respectively.
  Each subscale is calculated by obtaining the mean value of all of the answered items within the corresponding scale (possible value 0 to 4) and then multiplying by 25 to obtain the scale score (range 0 to 100).
Adherence | From enrollment to 16 weeks after SUPPORT program initiation
  To describe patient adherence to SUPPORT program at 8- and 16 weeks after SUPPORT program initiation.
  Adherence (at 8 weeks and 16 weeks after starting the program): How closely were you able to follow the SUPPORT program recommendations after starting the program? (Followed all recommendations; Followed most recommendations; Followed some recommendations; Rarely followed recommendations; Did not follow any recommendations).
Patient Satisfaction with the SUPPORT Program | From enrollment to 16 weeks after SUPPORT program initiation
  To describe patient satisfaction to SUPPORT program at 8- and 16 weeks after SUPPORT program initiation.
  Satisfaction (at 8 weeks after starting the program): How satisfied are you with the SUPPORT program? (Very satisfied; Satisfied; Neutral; Dissatisfied; Very dissatisfied).
PROMIS-57 - Patient Reported Outcomes Measurement Information System | From enrollment to 16 weeks after SUPPORT program initiation
  To compare anxiety, depression, fatigue, pain, physical function, sleep disturbance, and social roles using the NIH Patient Reported Outcomes Measurement Information System (PROMIS-57) profile at 8- and 16-weeks after SUPPORT program initiation.
  PROMIS-57 measures are scored on the T-score metric - in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. High scores mean more of the concept being measured (e.g., more Fatigue, more Physical Function).
Large Language Model usability (SUS - the System Usability Scale) | From enrollment to the end of treatment at 8 weeks
  To evaluate a large language model based digital coach's ability to be integrated into a self managed pelvic floor program. The System Usability Scale (SUS) is a 10-item questionnaire that provides a single composite score representing the overall usability of the system being evaluated. SUS scores range from 0 to 100, with higher scores indicating greater usability.
Attitudes toward Large Language Model Use (WAI-TECH-SF - Working Alliance Inventory for Online Interventions-Short Form) | From enrollment to the end of treatment at 8 weeks
  To assess patient satisfaction and attitudes toward use of a LLM as part of a self managed program. The Working Alliance Inventory for Online Interventions-Short Form (WAI-TECH-SF) is a 12-item self-report questionnaire that assess the therapeutic alliance between a patient and an online program. The scale ranges from 1 (never) to 5 (always). Higher scores indicate a stronger alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kenton, MD, Principal Investigator — University of Chicago; James Griffith, PhD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zoorob D, Higgins M, Swan K, Cummings J, Dominguez S, Carey E. Barriers to Pelvic Floor Physical Therapy Regarding Treatment of High-Tone Pelvic Floor Dysfunction. Female Pelvic Med Reconstr Surg. 2017 Nov/Dec;23(6):444-448. doi: 10.1097/SPV.0000000000000401. PMID 28145917
- [Background] Clason C, Sterner-Stein K, Hirschman KB, Barg FK, Riegel B. Developing effective health coaches: Experience gained in a clinical trial of a health coach intervention. Patient Educ Couns. 2023 Mar;108:107592. doi: 10.1016/j.pec.2022.107592. Epub 2022 Dec 9. PMID 36516655
- [Background] Al-Anezi FM. Exploring the use of ChatGPT as a virtual health coach for chronic disease management. Learn Health Syst. 2024 Jan 11;8(3):e10406. doi: 10.1002/lrh2.10406. eCollection 2024 Jul. PMID 39036525
- [Background] Hegde N, Vardhan M, Nathani D, Rosenzweig E, Speed C, Karthikesalingam A, Seneviratne M. Infusing behavior science into large language models for activity coaching. PLOS Digit Health. 2024 Apr 2;3(4):e0000431. doi: 10.1371/journal.pdig.0000431. eCollection 2024 Apr. PMID 38564502
- [Background] Stade EC, Stirman SW, Ungar LH, Boland CL, Schwartz HA, Yaden DB, Sedoc J, DeRubeis RJ, Willer R, Eichstaedt JC. Large language models could change the future of behavioral healthcare: a proposal for responsible development and evaluation. Npj Ment Health Res. 2024 Apr 2;3(1):12. doi: 10.1038/s44184-024-00056-z. PMID 38609507
- [Background] Wu JM, Vaughan CP, Goode PS, Redden DT, Burgio KL, Richter HE, Markland AD. Prevalence and trends of symptomatic pelvic floor disorders in U.S. women. Obstet Gynecol. 2014 Jan;123(1):141-148. doi: 10.1097/AOG.0000000000000057. PMID 24463674
- [Background] Yazdany T, Jakus-Waldman S, Jeppson PC, Schimpf MO, Yurteri-Kaplan LA, Ferzandi TR, Weber-LeBrun E, Knoepp L, Mamik M, Viswanathan M, Ward RM; American Urogynecologic Society. American Urogynecologic Society Systematic Review: The Impact of Weight Loss Intervention on Lower Urinary Tract Symptoms and Urinary Incontinence in Overweight and Obese Women. Female Pelvic Med Reconstr Surg. 2020 Jan/Feb;26(1):16-29. doi: 10.1097/SPV.0000000000000802. PMID 31860569
- [Background] Woodburn KL, Tran MC, Casas-Puig V, Ninivaggio CS, Ferrando CA. Compliance With Pelvic Floor Physical Therapy in Patients Diagnosed With High-Tone Pelvic Floor Disorders. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):94-97. doi: 10.1097/SPV.0000000000000732. PMID 31045618
- [Background] Sigurdardottir T, Steingrimsdottir T, Geirsson RT, Halldorsson TI, Aspelund T, Bo K. Can postpartum pelvic floor muscle training reduce urinary and anal incontinence?: An assessor-blinded randomized controlled trial. Am J Obstet Gynecol. 2020 Mar;222(3):247.e1-247.e8. doi: 10.1016/j.ajog.2019.09.011. Epub 2019 Sep 14. PMID 31526791
- [Background] Siddiqui NY, Ammarell N, Wu JM, Sandoval JS, Bosworth HB. Urinary Incontinence and Health-Seeking Behavior Among White, Black, and Latina Women. Female Pelvic Med Reconstr Surg. 2016 Sep-Oct;22(5):340-5. doi: 10.1097/SPV.0000000000000286. PMID 27171320
- [Background] Segal JL, Vassallo B, Kleeman S, Silva WA, Karram MM. Prevalence of persistent and de novo overactive bladder symptoms after the tension-free vaginal tape. Obstet Gynecol. 2004 Dec;104(6):1263-9. doi: 10.1097/01.AOG.0000147596.44421.72. PMID 15572487
- [Background] Rhodes RE, Fiala B. Building motivation and sustainability into the prescription and recommendations for physical activity and exercise therapy: the evidence. Physiother Theory Pract. 2009 Jul;25(5-6):424-41. doi: 10.1080/09593980902835344. PMID 19842866
- [Background] Markland AD, Richter HE, Fwu CW, Eggers P, Kusek JW. Prevalence and trends of urinary incontinence in adults in the United States, 2001 to 2008. J Urol. 2011 Aug;186(2):589-93. doi: 10.1016/j.juro.2011.03.114. PMID 21684555
- [Background] Mandimika CL, Murk W, Mcpencow AM, Lake AG, Miller D, Connell KA, Guess MK. Racial Disparities in Knowledge of Pelvic Floor Disorders Among Community-Dwelling Women. Female Pelvic Med Reconstr Surg. 2015 Sep-Oct;21(5):287-92. doi: 10.1097/SPV.0000000000000182. PMID 26313495
- [Background] Kotarinos RK. Pelvic floor physical therapy in urogynecologic disorders. Curr Womens Health Rep. 2003 Aug;3(4):334-9. PMID 12844459
- [Background] Kiyosaki K, Ackerman AL, Histed S, Sevilla C, Eilber K, Maliski S, Rogers RG, Anger J. Patients' understanding of pelvic floor disorders: what women want to know. Female Pelvic Med Reconstr Surg. 2012 May-Jun;18(3):137-42. doi: 10.1097/SPV.0b013e318254f09c. PMID 22543763
- [Background] Hatchett L, Hebert-Beirne J, Tenfelde S, Lavender MD, Brubaker L. Knowledge and perceptions of pelvic floor disorders among african american and latina women. Female Pelvic Med Reconstr Surg. 2011 Jul;17(4):190-4. doi: 10.1097/SPV.0b013e318229dd5c. PMID 22453850
- [Background] Harlow BL, Bavendam TG, Palmer MH, Brubaker L, Burgio KL, Lukacz ES, Miller JM, Mueller ER, Newman DK, Rickey LM, Sutcliffe S, Simons-Morton D. The Prevention of Lower Urinary Tract Symptoms (PLUS) Research Consortium: A Transdisciplinary Approach Toward Promoting Bladder Health and Preventing Lower Urinary Tract Symptoms in Women Across the Life Course. J Womens Health (Larchmt). 2018 Mar;27(3):283-289. doi: 10.1089/jwh.2017.6566. Epub 2017 Sep 15. PMID 29634445
- [Background] FitzGerald MP, Kotarinos R. Rehabilitation of the short pelvic floor. II: Treatment of the patient with the short pelvic floor. Int Urogynecol J Pelvic Floor Dysfunct. 2003 Oct;14(4):269-75; discussion 275. doi: 10.1007/s00192-003-1050-7. Epub 2003 Aug 7. PMID 14530840
- [Background] Felde G, Bjelland I, Hunskaar S. Anxiety and depression associated with incontinence in middle-aged women: a large Norwegian cross-sectional study. Int Urogynecol J. 2012 Mar;23(3):299-306. doi: 10.1007/s00192-011-1564-3. Epub 2011 Nov 9. PMID 22068320
- [Background] Dumoulin C, Hay-Smith EJ, Mac Habee-Seguin G. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2014 May 14;(5):CD005654. doi: 10.1002/14651858.CD005654.pub3. PMID 24823491
- [Background] Berger AA, Tan-Kim J, Menefee SA. Long-term Risk of Reoperation After Synthetic Mesh Midurethral Sling Surgery for Stress Urinary Incontinence. Obstet Gynecol. 2019 Nov;134(5):1047-1055. doi: 10.1097/AOG.0000000000003526. PMID 31599825
- [Background] Alewijnse D, Mesters I, Metsemakers J, van den Borne B. Predictors of long-term adherence to pelvic floor muscle exercise therapy among women with urinary incontinence. Health Educ Res. 2003 Oct;18(5):511-24. doi: 10.1093/her/cyf043. PMID 14572013
- [Background] Barber MD, Spino C, Janz NK, Brubaker L, Nygaard I, Nager CW, Wheeler TL; Pelvic Floor Disorders Network. The minimum important differences for the urinary scales of the Pelvic Floor Distress Inventory and Pelvic Floor Impact Questionnaire. Am J Obstet Gynecol. 2009 May;200(5):580.e1-7. doi: 10.1016/j.ajog.2009.02.007. PMID 19375574
- [Background] Alas AN, Dunivan GC, Wieslander CK, Sevilla C, Barrera B, Rashid R, Maliski S, Eilber K, Rogers RG, Anger JT. Health Care Disparities Among English-Speaking and Spanish-Speaking Women With Pelvic Organ Prolapse at Public and Private Hospitals: What Are the Barriers? Female Pelvic Med Reconstr Surg. 2016 Nov/Dec;22(6):460-466. doi: 10.1097/SPV.0000000000000315. PMID 27636216